CLINICAL TRIAL: NCT02576717
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Double-Dummy, Active Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of RPC1063 Administered Orally To Relapsing Multiple Sclerosis Patients
Brief Title: A Multi-Site, Open-Label Extension Trial of Oral RPC1063 in Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPC01-3001
Record Dates: First submitted 2015-09-28; First posted 2015-10-15 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: MS; RMS; Multiple Sclerosis; Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 mg RPC1063 (Ozanimod) oral capsule (Experimental): 1 mg RPC1063 (Ozanimod) oral capsule daily
  Interventions: Drug: RPC1063

INTERVENTIONS:
Drug: RPC1063
  Other Names: Ozanimod

SUMMARY:
The purpose of the trial is to determine the safety and efficacy of RPC1063 in patients with relapsing multiple sclerosis.

DETAILED DESCRIPTION:
The trial is an open label extension study. Eligible patients from the RPC01-201, RPC01-301, and RPC01-1001 trials diagnosed with relapsing Multiple Sclerosis (RMS) will be enrolled to receive study drug until the end of the trial or until the Sponsor discontinues the development program.

ELIGIBILITY:
Eligibility Criteria:

To be eligible to participate in this trial, patients must meet all of the following criteria:

1. Completed one of the parent trials
2. Does not have a condition that would require withdrawal from one of the parent trials
3. Has no conditions requiring treatment with a prohibited concomitant medication
4. Is not receiving treatment with any of the following drugs or interventions within the corresponding timeframe:

   At Baseline (Day 1)
   * CYP2C8 inhibitors (eg, gemfibrozil or clopidogrel) or inducers (eg, rifampicin) Two weeks prior to Baseline (Day 1)
   * Monoamine oxidase inhibitors (eg, selegiline, phenelzine)
5. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments
6. Female patients of childbearing potential:

Must agree to practice a highly effective method of contraception throughout the study until completion of the 90-day Safety Follow-up Visit. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly.

Acceptable methods of birth control in this study are the following:

* Combined hormonal (estrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, or implantable
* Placement of an intrauterine device (IUD)
* Placement of an intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomised partner
* Sexual abstinence.

Exclusion Criteria:

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2494 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (175):
- United States (19):
  - Local Institution - 115, Phoenix, Arizona
  - Local Institution - 118, Phoenix, Arizona
  - Local Institution - 110, Berkeley, California
  - Local Institution - 103, Fresno, California
  - Local Institution - 122, Long Beach, California
  - Local Institution - 112, Sacramento, California
  - Local Institution - 120, San Francisco, California
  - Local Institution - 114, Maitland, Florida
  - Local Institution - 123, Port Charlotte, Florida
  - Local Institution - 124, Sunrise, Florida
  - Local Institution - 147, Tampa, Florida
  - Local Institution - 137, Golden Valley, Minnesota
  - Local Institution - 170, Las Vegas, Nevada
  - Local Institution - 143, Raleigh, North Carolina
  - Local Institution - 107, Westerville, Ohio
  - Local Institution - 144, Knoxville, Tennessee
  - Local Institution - 138, Lubbock, Texas
  - Local Institution - 179, Round Rock, Texas
  - Local Institution - 141, Kirkland, Washington
- Belarus (7):
  - Local Institution - 907, Grodno
  - Local Institution - 904, Homyel
  - Local Institution - 902, Minsk
  - Local Institution - 901, Minsk
  - Local Institution - 903, Minsk
  - Local Institution - 905, Vitebsk
  - Local Institution - 906, Vitebsk
- Belgium (3):
  - Local Institution - 256, Bruges
  - Local Institution - 255, Brussels
  - Local Institution - 252, Montegnée
- Bosnia and Herzegovina (2):
  - Local Institution - 913, Banja Luka
  - Local Institution - 911, Sarajevo
- Bulgaria (7):
  - Local Institution - 453, Sofia
  - Local Institution - 454, Sofia
  - Local Institution - 452, Sofia
  - Local Institution - 456, Sofia
  - Local Institution - 457, Sofia
  - Local Institution - 460, Sofia
  - Local Institution - 455, Sofia
- Croatia (4):
  - Local Institution - 923, Osijek
  - Local Institution - 921, Zagreb
  - Local Institution - 922, Zagreb
  - Local Institution - 924, Zagreb
- Estonia (3):
  - Local Institution - 473, Tallinn
  - Local Institution - 471, Tallinn
  - Local Institution - 472, Tartu
- Georgia (5):
  - Local Institution - 301, Tbilisi
  - Local Institution - 302, Tbilisi
  - Local Institution - 304, Tbilisi
  - Local Institution - 306, Tbilisi
  - Local Institution - 303, Tbilisi
- Germany (3):
  - Local Institution - 487, Leipzig
  - Local Institution - 496, Potsdam
  - Local Institution - 488, Ulm
- Greece (4):
  - Local Institution - 552, Athens
  - Local Institution - 553, Athens
  - Local Institution - 551, Athens
  - Local Institution - 555, Thessaloniki
- Hungary (5):
  - Local Institution - 352, Budapest
  - Local Institution - 356, Budapest
  - Local Institution - 354, Esztergom
  - Local Institution - 358, Kistarcsa
  - Local Institution - 351, Nyíregyháza
- Italy (5):
  - Local Institution - 654, Catania
  - Local Institution - 653, Cefalù
  - Local Institution - 655, Milan
  - Local Institution - 659, Montichiari
  - Local Institution - 651, Roma
- Latvia (2):
  - Local Institution - 562, Riga
  - Local Institution - 561, Riga
- Lithuania (2):
  - Local Institution - 622, Kaunas, Kaunas County
  - Local Institution - 621, Klaipėda
- Moldova (3):
  - Local Institution - 932, Chisinau
  - Local Institution - 931, Chisinau
  - Local Institution - 933, Chisinau
- New Zealand (2):
  - Local Institution - 511, Christchurch
  - Local Institution - 510, Hamilton
- Poland (32):
  - Local Institution - 434, Warsaw, Masovian Voivodeship
  - Local Institution - 401, Bialystok
  - Local Institution - 423, Bydgoszcz
  - Local Institution - 406, Czeladź
  - Local Institution - 405, Gdansk
  - Local Institution - 432, Jarosław
  - Local Institution - 417, Katowice
  - Local Institution - 427, Katowice
  - Local Institution - 426, Katowice
  - Local Institution - 407, Katowice
  - Local Institution - 424, Kielce
  - Local Institution - 404, Konstancin-Jeziorna
  - Local Institution - 414, Krakow
  - Local Institution - 411, Lódzkie
  - Local Institution - 429, Lublin
  - Local Institution - 412, Lublin
  - Local Institution - 420, Lublin
  - Local Institution - 431, Mazowieckie
  - Local Institution - 415, Olsztyn
  - Local Institution - 421, Plewiska
  - Local Institution - 425, Pomorskie
  - Local Institution - 408, Poznan
  - Local Institution - 418, Poznan
  - Local Institution - 433, Rybnik
  - Local Institution - 435, Rzeszów
  - Local Institution - 419, Szczecin
  - Local Institution - 402, Warminsko-mazurskie
  - Local Institution - 410, Warsaw
  - Local Institution - 428, Warsaw
  - Local Institution - 422, Warsaw
  - Local Institution - 403, Warsaw
  - Local Institution - 413, Warsaw
- Portugal (3):
  - Local Institution - 772, Braga
  - Local Institution - 775, Coimbra
  - Local Institution - 773, Torres Vedras
- Romania (9):
  - Local Institution - 503, Brasov
  - Local Institution - 509, Bucharest
  - Local Institution - 504, Bucharest
  - Local Institution - 520, Bucharest
  - Local Institution - 502, Campulung Muscel
  - Local Institution - 508, Cluj-Napoca
  - Local Institution - 501, Cluj-Napoca
  - Local Institution - 507, Constanța
  - Local Institution - 506, Timișoara
- Serbia (6):
  - Local Institution - 602, Belgrade
  - Local Institution - 603, Belgrade
  - Local Institution - 604, Belgrade
  - Local Institution - 601, Belgrade
  - Local Institution - 605, Kragujevac
  - Local Institution - 606, Niš
- Slovakia (3):
  - Local Institution - 946, Bratislava
  - Local Institution - 942, Lučenec
  - Local Institution - 945, Trnava
- Local Institution - 953, Pretoria, South Africa
- Spain (12):
  - Local Institution - 756, Barcelona
  - Local Institution - 758, Barcelona
  - Local Institution - 761, Bilbao
  - Local Institution - 759, Donostia / San Sebastian
  - Local Institution - 760, Girona
  - Local Institution - 757, Madrid
  - Local Institution - 754, Majadahonda
  - Local Institution - 764, Pamplona/ Navarra
  - Local Institution - 766, Sant Joan Despí
  - Local Institution - 755, Sevillla
  - Local Institution - 767, Valencia
  - Local Institution - 752, Valencia
- Local Institution - 780, Gothenburg, Sweden
- Ukraine (29):
  - Local Institution - 823, Cherkasy
  - Local Institution - 830, Chernihiv
  - Local Institution - 805, Chernihiv
  - Local Institution - 813, Chernivtsi
  - Local Institution - 802, Dnipropetrovsk
  - Local Institution - 815, Dnipropetrovsk
  - Local Institution - 801, Ivano-Frankivsk
  - Local Institution - 829, Ivano-Frankivsk
  - Local Institution - 814, Kharkiv
  - Local Institution - 827, Kharkiv
  - Local Institution - 832, Kharkiv
  - Local Institution - 811, Kherson
  - Local Institution - 822, Kyiv
  - Local Institution - 803, Kyiv
  - Local Institution - 818, Kyiv
  - Local Institution - 824, Kyiv
  - Local Institution - 817, Lutsk
  - Local Institution - 812, Lviv
  - Local Institution - 821, Lviv
  - Local Institution - 810, Odesa
  - Local Institution - 831, Odesa
  - Local Institution - 804, Odesa
  - Local Institution - 826, Poltava
  - Local Institution - 820, Uzhhorod
  - Local Institution - 809, Vinnytsia
  - Local Institution - 825, Zaporizhia
  - Local Institution - 828, Zaporizhzhia
  - Local Institution - 806, Zaporizhzhya
  - Local Institution - 819, Zhytomyr
- United Kingdom (3):
  - Local Institution - 965, East Sussex
  - Local Institution - 963, Inverness
  - Local Institution - 964, Sheffield

REFERENCES:
- [Derived] Selmaj KW, Steinman L, Comi G, Bar-Or A, Arnold DL, Hartung HP, Montalban X, Havrdova EK, Sheffield JK, Krakovich A, Cheng CY, Riolo JV, Pachai C, Thorpe A, DeBoer E, Kappos L, Cohen JA, Cree BA. Long-term safety and efficacy of ozanimod in relapsing multiple sclerosis: Final analysis of the DAYBREAK open-label extension trial. Mult Scler. 2025 Nov;31(13):1557-1571. doi: 10.1177/13524585251382796. Epub 2025 Nov 5. PMID 41190505
- [Derived] Cohen JA, Arnold DL, DeLuca J, Hartung HP, Kappos L, Comi G, Selmaj K, Steinman L, Bar-Or A, Montalban X, Havrdova EK, Sheffield JK, Pachai C, Cheng CY, Riolo JV, Cree BA. Brain atrophy and associations with long-term disability and cognitive function in participants with relapsing multiple sclerosis treated with ozanimod: Results from phase 3 and open-label extension trials. Mult Scler. 2025 Sep;31(10):1218-1230. doi: 10.1177/13524585251355842. Epub 2025 Jul 23. PMID 40698614
- [Derived] Regueiro M, Siegmund B, Horst S, Moslin R, Charles L, Petersen A, Tatosian D, Wu H, Lawlor G, Fischer M, D'Haens G, Colombel JF. Concomitant Administration of Ozanimod and Serotonergic Antidepressants in Patients With Ulcerative Colitis or Relapsing Multiple Sclerosis. Inflamm Bowel Dis. 2025 Apr 10;31(4):1010-1017. doi: 10.1093/ibd/izae136. PMID 39018016
- [Derived] Naismith RT, Cohen JA, Bar-Or A, Comi G, Selmaj KW, Hartung HP, Sheffield JK, Krakovich A, Tatosian D, Cheng CY, Reardon J, Khaychuk V, Riolo JV, Silva D, Cree BA. Concurrent administration of serotonergic antidepressants and ozanimod in participants with relapsing multiple sclerosis from the open-label extension DAYBREAK trial. Mult Scler. 2024 Feb;30(2):177-183. doi: 10.1177/13524585231216854. Epub 2023 Dec 21. PMID 38130041
- [Derived] Cree BAC, Maddux R, Bar-Or A, Hartung HP, Kaur A, Brown E, Li Y, Hu Y, Sheffield JK, Silva D, Harris S. SARS-CoV-2 vaccination and infection in ozanimod-treated participants with relapsing multiple sclerosis. Ann Clin Transl Neurol. 2023 Oct;10(10):1725-1737. doi: 10.1002/acn3.51862. Epub 2023 Aug 7. PMID 37550942
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have participated in Trial RPC01-201, Trial RPC01-301, and/or Trial RPC01-1001 prior to joining RPC01-3001.
Pre-assignment Details: Participants were Pooled According to Treatment Assignment in Parent Trial. A total of 2494 participants were treated, however, in the parent treatment groups 3 participants planned for IFN β-1a received RPC1063 0.5 mg, 1 participant planned for IFN β 1a received RPC1063 1 mg, and 1 participant planned for ozanimod 0.5 mg received RPC1063 1 mg. The parent placebo 0.5 mg and 1 mg study groups were consolidated into the 0.5 mg and 1 mg RPC1063 groups.
Groups:
- Parent Treatment Group IFN-B-1a 30 ug; Parent Treatment Group: RPC1063 0.5 mg; Parent Treatment Group: RPC1063 1.0 mg: Participants received a 7-day titration regimen of RPC1063, as applicable to reach the targeted dose of 1.0 mg which was taken by mouth once per day until the end of the trial or until the Sponsor discontinued the development program. Participants were instructed to take RPC1063 at approximately the same time each day with or without food.
Period: Overall Study
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Started (Started = ITT Participants were included in the treatment group based on the planned treatment (received at randomization) in the parent study.) | 740 | 875 | 879
Transferred From IFN β-1a Parent Group | 0 | 3 (Participants were planned for IFN β-1a received RPC1063 0.5 mg) | 1 (Participant was planned for IFN β 1a but received RPC1063 1 mg)
Transferred From RPC1063 0.5 mg Parent Group | 0 | 0 | 1 (Participant was planned for RPC1063 0.5 mg but received RPC1063 1 mg)
Randomized to Placebo in the Parent Study | 0 | 37 | 35
Safety Population (Participants were included in the treatment group based on the treatment that they actually received in the parent study.) | 736 | 877 | 881
Completed | 564 | 691 | 695
Not Completed | 176 | 184 | 184
Not completed — Other Reasons | 16 | 18 | 15
Not completed — Covid-19 Pandemic | 0 | 1 | 1
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Physician Decision | 3 | 8 | 9
Not completed — Participant Voluntarily Withdrew from Study | 91 | 82 | 85
Not completed — Death | 3 | 5 | 3
Not completed — Lost to Follow-up | 9 | 10 | 19
Not completed — Protocol Violation | 4 | 0 | 5
Not completed — Lack of Efficacy | 24 | 28 | 20
Not completed — Adverse Event | 26 | 32 | 26

BASELINE CHARACTERISTICS:
Population: Demographics were summarized using the safety population - all participants enrolled in study RPC01-3001 who received at least one dose of open-label RPC1063.
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg | Total
Number analyzed (Participants) | 736 | 877 | 881 | 2494
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 736 | 877 | 881 | 2494
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 498 | 595 | 575 | 1668
  Male | 238 | 282 | 306 | 826
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 16 | 27
  Not Hispanic or Latino | 733 | 869 | 865 | 2467
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 734 | 865 | 875 | 2474
    Black or African American | 1 | 7 | 6 | 14
    Asian | 0 | 3 | 0 | 3
    Other | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporarily associated with the use of medicinal product, whether or not considered related to the investigational medicinal product.
Time Frame: From first dose to 90-days post last dose (an average of 65 months up to a max of 85 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Participants | 668 | 775 | 776

2. Primary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose to 90-days post last dose (an average of 65 months up to a max of 85 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Participants | 108 | 139 | 134

3. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: as for outcome 1
Time Frame: From first dose to 90-days post last dose (an average of 65 months up to a max of 85 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Participants | 35 | 35 | 28

4. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Withdrawal
Description: as for outcome 1
Time Frame: From first dose to 90-days post last dose (an average of 65 months up to a max of 85 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Participants | 32 | 35 | 28

5. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) of Special Interest
Description: as for outcome 1
Time Frame: From first dose to 90-days post last dose (an average of 65 months up to a max of 85 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Participants
  Infections and infestations | 19 | 26 | 19
  Neoplasms benign, malignant and unspecified (Incl cysts and polyps) | 9 | 14 | 16
  Blood and lymphatic system disorders | 0 | 0 | 1
  Nervous system disorders | 0 | 2 | 1
  Eye disorders | 5 | 2 | 2
  Cardiac disorders | 0 | 1 | 2
  Hepatobiliary disorders | 0 | 1 | 0
  Skin and subcutaneous tissue disorders | 0 | 0 | 1
  Congenital, familial and genetic disorders | 1 | 0 | 0
  Investigations | 15 | 14 | 8

6. Primary Outcome: Number of Participants With Abnormalities in Blood Absolute Lymphocyte Count (ALC)
Description: An absolute lymphocyte count (ALC) is a part of a blood test that measures the number of lymphocytes, a type of white blood cell, in the blood. Lymphocytes help fight infections and diseases. Reductions in ALC levels for participants in this study is expected and is a primary pharmacodynamic effect of RPC1063.
  LLN = Lower limit of normal
Time Frame: From first dose up until last dose of study treatment (up to approximately 82 months)
Population: All treated participants with at least one on treatment ALC assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 727 | 868 | 877
Participants
  ALC < 0.2 x 10^9/L | 33 | 33 | 27
  ALC < 0.5 x 10^9/L | 265 | 323 | 339
  ALC < 0.8 x 10^9/L | 497 | 620 | 616
  ALC < LLN | 592 | 703 | 704

7. Primary Outcome: Number of Participants With Abnormalities in White Blood Cell Count (WBC)
Description: A white blood cell count is a part of a blood test that measures the number of white blood cells in the blood. White blood cells help fight infections and diseases.
  LLN = Lower limit of normal
Time Frame: From first dose up until last dose of study treatment (up to approximately 82 months)
Population: All treated participants with at least one on treatment WBC assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 727 | 868 | 877
Participants
  Total WBC > 20 x 10^9/L | 0 | 0 | 2
  Total WBC < 3 x 10^9/L | 27 | 48 | 43
  Total WBC < 2 x 10^9/L | 0 | 2 | 0
  Total WBC < 1 x 10^9/L | 0 | 0 | 0
  Total WBC < LLN | 92 | 107 | 108

8. Primary Outcome: Number of Participants With Abnormalities in Blood Absolute Neutrophil Count (ANC)
Description: An absolute neutrophil count is a part of a blood test that measures the number of neutrophils, a type of white blood cell, in the blood. Neutrophils help fight infections and diseases.
Time Frame: From first dose up until last dose of study treatment (up to approximately 82 months)
Population: All treated participants with at least one on treatment ANC assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 727 | 868 | 877
Participants | 0 | 2 | 1

9. Primary Outcome: Number of Participants With Abnormalities in Specific Liver Function Tests
Description: The number of participants with laboratory abnormalities in specific liver tests above ULN by category. ULN = Upper Limit of Normal
Time Frame: From first dose up until last dose of study treatment (up to approximately 82 months)
Population: All treated participants with at least one on treatment liver function test
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 734 | 875 | 880
Participants
  > 1 x ULN | 311 | 353 | 353
  >= 2 x ULN | 90 | 100 | 107
  >= 3 x ULN | 32 | 30 | 29
  >= 4 x ULN | 16 | 19 | 6
  >= 5 x ULN | 8 | 12 | 0
  >= 10 x ULN | 4 | 5 | 0

10. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Result Abnormalities
Description: An electrocardiogram (ECG) measures electrical activity of the heart to detect cardiac problems.
Time Frame: From first dose to 28-days post last dose (an average of 63 months up to a max of 83 months)
Population: All treated participants with baseline and at least one post baseline ECG assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 876 | 880
Participants
  QT > 480 (ms) | 6 | 5 | 3
  QT > 500 (ms) | 1 | 0 | 0
  QTcF > 450 (ms) | 44 | 49 | 44
  QTcF > 480 (ms) | 1 | 5 | 3
  QTcF > 500 (ms) | 0 | 0 | 0
  QTcB > 450 (ms) | 173 | 186 | 184
  QTcB > 480 (ms) | 8 | 15 | 13
  QTcB > 500 (ms) | 0 | 2 | 0
  Change from Baseline in QTcF >30 ms | 134 | 140 | 120
  Change from Baseline in QTcF >60 ms | 0 | 5 | 6
  Change from Baseline in QTcB >30 ms | 183 | 215 | 205
  Change from Baseline in QTcB >60 ms | 5 | 9 | 13
  Atrial Ventricular Bock or Conduction Ratio, 2:1 | 0 | 0 | 1

11. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Vital Signs
Description: Vital signs included body temperature, sitting heart rate/pulse (HR), sitting systolic blood pressure (SBP), sitting diastolic blood pressure (DBP).
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and 60 months after first dose of study therapy
Population: All treated participants with baseline and on study assessment for that vital sign at 60 months post first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 567 | 715 | 707
Participants
  Temperature (C) >38.5 and an increase from Baseline of at least 1: number analyzed (Participants) | 566 | 715 | 707
  Temperature (C) >38.5 and an increase from Baseline of at least 1 | 0 | 0 | 0
  Heart Rate (bpm) >120 beats per minute post-Baseline or an increase from Baseline of >20 bpm: number analyzed (Participants) | 567 | 715 | 706
  Heart Rate (bpm) >120 beats per minute post-Baseline or an increase from Baseline of >20 bpm | 15 | 19 | 26
  Heart Rate (bpm) >120 bpm post-Baseline if Baseline <=120 bpm: number analyzed (Participants) | 567 | 715 | 706
  Heart Rate (bpm) >120 bpm post-Baseline if Baseline <=120 bpm | 0 | 0 | 0
  Heart Rate (bpm) An increase from Baseline of more than 20 bpm: number analyzed (Participants) | 567 | 715 | 706
  Heart Rate (bpm) An increase from Baseline of more than 20 bpm | 15 | 19 | 26
  Heart Rate (bpm) <45 bpm post-Baseline or a decrease from Baseline of more than 20bpm: number analyzed (Participants) | 567 | 715 | 706
  Heart Rate (bpm) <45 bpm post-Baseline or a decrease from Baseline of more than 20bpm | 7 | 12 | 8
  Heart Rate (bpm) <45 bpm post-Baseline if Baseline >=45 bpm: number analyzed (Participants) | 567 | 715 | 706
  Heart Rate (bpm) <45 bpm post-Baseline if Baseline >=45 bpm | 0 | 0 | 0
  Heart Rate (bpm) A decrease from Baseline of more than 20 bpm: number analyzed (Participants) | 567 | 715 | 706
  Heart Rate (bpm) A decrease from Baseline of more than 20 bpm | 7 | 12 | 8
  Systolic Blood Pressure (mmHg) >180 mmHg post-Baseline or an increase from Baseline of >40 mmHg | 3 | 5 | 5
  Systolic Blood Pressure (mmHg) >180 mmHg post-Baseline if Baseline <=180 mmHg | 0 | 0 | 0
  Systolic Blood Pressure (mmHg) An increase from Baseline of more than 40 mmHg | 3 | 5 | 5
  Systolic Blood Pressure (mmHg) <90 mmHg post-Baseline or a decrease from Baseline >30 mmHg | 3 | 1 | 3
  Systolic Blood Pressure (mmHg) <90 mmHg post-Baseline if Baseline >=90 mmHg | 1 | 0 | 0
  Systolic Blood Pressure (mmHg) A decrease from Baseline of more than 30 mmHg | 2 | 1 | 3
  Diastolic Blood Pressure (mmHg) >105 mmHg post-Baseline or an increase from Baseline >30 mmHg | 2 | 4 | 4
  Diastolic Blood Pressure (mmHg) >105 mmHg post-Baseline if Baseline <=105 mmHg | 1 | 2 | 3
  Diastolic Blood Pressure (mmHg) An increase from Baseline of more than 30 mmHg | 1 | 2 | 2
  Diastolic Blood Pressure (mmHg) <50 mmHg post-Baseline or a decrease from Baseline of >30 mmHg | 1 | 2 | 0
  Diastolic Blood Pressure (mmHg) <50 mmHg post-Baseline if Baseline >=50 mmHg | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) A decrease from Baseline of more than 30 mmHg | 1 | 2 | 0

12. Primary Outcome: Number of Participants With Physical Examination Abnormalities
Description: The number of participants with abnormal physical examination results. The assessments included abdominal, extremity, head, heart, lungs, neck, neurological non-MS, other and skin assessments.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 84 months post first dose.
Population: All treated participants with baseline and at least one on treatment physical assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Participants
  Baseline - Abdominal | 0 | 0 | 1
  Baseline - Extremities | 3 | 2 | 8
  Baseline - Head | 0 | 1 | 1
  Baseline - Heart | 1 | 0 | 1
  Baseline - Lungs | 0 | 1 | 2
  Baseline - Neck | 0 | 1 | 3
  Baseline - Neurological-Non-MS | 1 | 1 | 5
  Baseline - Other | 2 | 6 | 4
  Baseline - Skin | 17 | 17 | 16
  Month 12 - Abdominal: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Abdominal | 1 | 2 | 2
  Month 12 - Extremities: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Extremities | 2 | 4 | 6
  Month 12 - Head: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Head | 2 | 2 | 3
  Month 12 - Heart: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Heart | 3 | 0 | 0
  Month 12 - Lungs: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Lungs | 0 | 0 | 1
  Month 12 - Neck: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Neck | 0 | 1 | 3
  Month 12 - Neurological-Non-MS: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Neurological-Non-MS | 1 | 3 | 0
  Month 12 - Other: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Other | 2 | 4 | 2
  Month 12 - Skin: number analyzed (Participants) | 708 | 848 | 854
  Month 12 - Skin | 25 | 24 | 21
  Month 24 - Abdominal: number analyzed (Participants) | 684 | 811 | 831
  Month 24 - Abdominal | 0 | 2 | 2
  Month 24 -Extremities: number analyzed (Participants) | 684 | 811 | 831
  Month 24 -Extremities | 5 | 9 | 6
  Month 24 - Head: number analyzed (Participants) | 684 | 811 | 831
  Month 24 - Head | 3 | 4 | 2
  Month 24 - Lungs: number analyzed (Participants) | 684 | 811 | 831
  Month 24 - Lungs | 0 | 1 | 3
  Month 24 - Neck: number analyzed (Participants) | 684 | 811 | 831
  Month 24 - Neck | 1 | 1 | 2
  Month 24 - Neurological-Non-MS: number analyzed (Participants) | 684 | 811 | 831
  Month 24 - Neurological-Non-MS | 2 | 1 | 3
  Month 24 - Other: number analyzed (Participants) | 684 | 811 | 831
  Month 24 - Other | 2 | 3 | 3
  Month 24 - Skin: number analyzed (Participants) | 684 | 811 | 831
  Month 24 - Skin | 20 | 21 | 23
  Month 36 - Abdominal: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Abdominal | 1 | 1 | 1
  Month 36 - Extremities: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Extremities | 5 | 5 | 7
  Month 36 - Head: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Head | 1 | 0 | 4
  Month 36 - Heart: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Heart | 0 | 0 | 1
  Month 36 - Lungs: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Lungs | 1 | 2 | 1
  Month 36 - Neck: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Neck | 1 | 1 | 0
  Month 36 - Neurological-Non-MS: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Neurological-Non-MS | 1 | 1 | 4
  Month 36 - Other: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Other | 4 | 4 | 4
  Month 36 - Skin: number analyzed (Participants) | 640 | 774 | 794
  Month 36 - Skin | 22 | 32 | 34
  Month 48 - Abdominal: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Abdominal | 0 | 0 | 1
  Month 48 - Extremities: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Extremities | 4 | 7 | 5
  Month 48 - Head: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Head | 1 | 2 | 1
  Month 48 - Heart: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Heart | 0 | 0 | 1
  Month 48 - Lungs: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Lungs | 0 | 1 | 2
  Month 48 - Neck: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Neck | 0 | 1 | 0
  Month 48 - Neurological-Non-MS: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Neurological-Non-MS | 3 | 1 | 0
  Month 48 - Other: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Other | 2 | 3 | 4
  Month 48 - Skin: number analyzed (Participants) | 603 | 736 | 743
  Month 48 - Skin | 19 | 23 | 18
  Month 60 - Abdominal: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Abdominal | 1 | 2 | 0
  Month 60 - Extremities: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Extremities | 4 | 9 | 11
  Month 60 - Head: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Head | 1 | 1 | 1
  Month 60 - Heart: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Heart | 0 | 0 | 2
  Month 60 - Lungs: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Lungs | 0 | 1 | 2
  Month 60 - Neck: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Neck | 2 | 0 | 0
  Month 60 - Neurological-Non-MS: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Neurological-Non-MS | 2 | 1 | 4
  Month 60 - Other: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Other | 3 | 4 | 1
  Month 60 - Skin: number analyzed (Participants) | 580 | 717 | 718
  Month 60 - Skin | 16 | 28 | 18
  Month 72 - Abdominal: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Abdominal | 1 | 2 | 2
  Month 72 - Extremities: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Extremities | 4 | 5 | 5
  Month 72 - Head: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Head | 0 | 1 | 1
  Month 72 - Heart: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Heart | 0 | 0 | 0
  Month 72 - Lungs: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Lungs | 0 | 0 | 1
  Month 72 - Neck: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Neck | 1 | 0 | 0
  Month 72 - Neurological-Non-MS: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Neurological-Non-MS | 2 | 2 | 2
  Month 72 - Other: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Other | 5 | 3 | 2
  Month 72 - Skin: number analyzed (Participants) | 445 | 564 | 584
  Month 72 - Skin | 8 | 19 | 10
  Month 84 - Abdominal: number analyzed (Participants) | 0 | 7 | 10
  Month 84 - Abdominal |  | 1 | 0
  Month 84 - Extremities: number analyzed (Participants) | 0 | 7 | 10
  Month 84 - Extremities |  | 1 | 1
  Month 84 - Skin: number analyzed (Participants) | 0 | 7 | 10
  Month 84 - Skin |  | 2 | 0

13. Primary Outcome: Number of Participants Self-Identifying Suicidality by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a unique suicide risk assessment tool that supports suicide risk assessment through a series of simple, plain-language questions. The answers help users identify whether someone is at risk for suicide, assess the severity and immediacy of that risk, and gauge the level of support that the person needs.
  Results are displayed as the number of participants who answered "Yes" to at least one of the 10 questions in the suicidal ideation or suicidal behavior section.
  Ideation from 1 (wishing to be dead) - 5 (Active suicidal ideation with specific plan and intent) Behavior from 6 (Preparatory acts or behavior) - 10 (Completed suicide). Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 3 months thereafter up until 78 months post first dose.
Population: All treated participants with an assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 733 | 874 | 879
Participants
  At baseline (Suicidal Ideation or Behavior): number analyzed (Participants) | 393 | 431 | 417
  At baseline (Suicidal Ideation or Behavior) | 0 | 2 | 0
  At month 3 (Suicidal Ideation or Behavior) | 2 | 1 | 1
  At month 6 (Suicidal Ideation or Behavior): number analyzed (Participants) | 727 | 865 | 874
  At month 6 (Suicidal Ideation or Behavior) | 1 | 1 | 2
  At month 9 (Suicidal Ideation or Behavior): number analyzed (Participants) | 719 | 854 | 860
  At month 9 (Suicidal Ideation or Behavior) | 3 | 0 | 1
  At month 12 (Suicidal Ideation or Behavior): number analyzed (Participants) | 705 | 848 | 854
  At month 12 (Suicidal Ideation or Behavior) | 3 | 0 | 2
  At month 15 (Suicidal Ideation or Behavior): number analyzed (Participants) | 698 | 831 | 847
  At month 15 (Suicidal Ideation or Behavior) | 0 | 0 | 1
  At month 18 (Suicidal Ideation or Behavior): number analyzed (Participants) | 690 | 822 | 842
  At month 18 (Suicidal Ideation or Behavior) | 1 | 1 | 2
  At month 21 (Suicidal Ideation or Behavior): number analyzed (Participants) | 682 | 815 | 833
  At month 21 (Suicidal Ideation or Behavior) | 1 | 0 | 1
  At month 24 (Suicidal Ideation or Behavior): number analyzed (Participants) | 676 | 800 | 820
  At month 24 (Suicidal Ideation or Behavior) | 1 | 2 | 1
  At month 27 (Suicidal Ideation or Behavior): number analyzed (Participants) | 663 | 791 | 812
  At month 27 (Suicidal Ideation or Behavior) | 0 | 0 | 0
  At month 33 (Suicidal Ideation or Behavior): number analyzed (Participants) | 646 | 780 | 796
  At month 33 (Suicidal Ideation or Behavior) | 1 | 0 | 0
  At month 36 (Suicidal Ideation or Behavior): number analyzed (Participants) | 631 | 772 | 787
  At month 36 (Suicidal Ideation or Behavior) | 2 | 1 | 0
  At month 39 (Suicidal Ideation or Behavior): number analyzed (Participants) | 623 | 761 | 776
  At month 39 (Suicidal Ideation or Behavior) | 0 | 1 | 0
  At month 42 (Suicidal Ideation or Behavior): number analyzed (Participants) | 611 | 750 | 755
  At month 42 (Suicidal Ideation or Behavior) | 0 | 0 | 1
  At month 45 (Suicidal Ideation or Behavior): number analyzed (Participants) | 564 | 704 | 705
  At month 45 (Suicidal Ideation or Behavior) | 0 | 0 | 0
  At month 48 (Suicidal Ideation or Behavior): number analyzed (Participants) | 606 | 731 | 740
  At month 48 (Suicidal Ideation or Behavior) | 2 | 0 | 1
  At month 54 (Suicidal Ideation or Behavior): number analyzed (Participants) | 573 | 714 | 718
  At month 54 (Suicidal Ideation or Behavior) | 1 | 0 | 1
  At month 57 (Suicidal Ideation or Behavior): number analyzed (Participants) | 40 | 92 | 90
  At month 57 (Suicidal Ideation or Behavior) | 0 | 0 | 0
  At month 60 (Suicidal Ideation or Behavior): number analyzed (Participants) | 570 | 716 | 708
  At month 60 (Suicidal Ideation or Behavior) | 2 | 1 | 1
  At month 66 (Suicidal Ideation or Behavior): number analyzed (Participants) | 538 | 670 | 677
  At month 66 (Suicidal Ideation or Behavior) | 1 | 2 | 1
  At month 69 (Suicidal Ideation or Behavior): number analyzed (Participants) | 393 | 419 | 403
  At month 69 (Suicidal Ideation or Behavior) | 1 | 0 | 1
  At month 72 (Suicidal Ideation or Behavior): number analyzed (Participants) | 267 | 361 | 352
  At month 72 (Suicidal Ideation or Behavior) | 1 | 0 | 1
  At month 78 (Suicidal Ideation or Behavior): number analyzed (Participants) | 9 | 65 | 72
  At month 78 (Suicidal Ideation or Behavior) | 0 | 0 | 1

14. Primary Outcome: Number of Participants With Changes in Suicidality From Last Day on Treatment Per the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a unique suicide risk assessment tool that supports suicide risk assessment through a series of simple, plain-language questions. The answers help users identify whether someone is at risk for suicide, assess the severity and immediacy of that risk, and gauge the level of support that the person needs.
  Results are displayed as the number of participants who answered "Yes" to at least one of the 10 questions in the suicidal ideation or suicidal behavior section.
  Ideation from 1 (wishing to be dead) - 5 (Active suicidal ideation with specific plan and intent) Behavior from 6 (Preparatory acts or behavior) - 10 (Completed suicide).
Time Frame: 1, 4, 7, 14, 21, 28, and 90 days post last dose.
Population: All treated participants who discontinued study treatment and had at least one on study and one post-dose assessment. Prespecified to be collected in combination for all three study arms.
Measure: Count of Participants; unit: Participants
Groups:
- Combined Parent Treatment Group: Participants received a 7-day titration regimen of RPC1063, as applicable to reach the targeted dose of 1.0 mg which was taken by mouth once per day until the end of the trial or until the Sponsor discontinued the development program. Participants were instructed to take RPC1063 at approximately the same time each day with or without food.
Arm/Group | Combined Parent Treatment Group
Number analyzed (Participants) | 250
Participants
  End of Treatment | 3
  Follow-up Visit Day 1: number analyzed (Participants) | 96
  Follow-up Visit Day 1 | 0
  Follow-up Visit Day 4: number analyzed (Participants) | 99
  Follow-up Visit Day 4 | 0
  Follow-up Visit Day 7: number analyzed (Participants) | 99
  Follow-up Visit Day 7 | 0
  Follow-up Visit Day 14: number analyzed (Participants) | 99
  Follow-up Visit Day 14 | 0
  Follow-up Visit Day 21: number analyzed (Participants) | 91
  Follow-up Visit Day 21 | 0
  Safety Follow-up Visit (Day 28): number analyzed (Participants) | 219
  Safety Follow-up Visit (Day 28) | 0
  Follow-up Visit Day 90: number analyzed (Participants) | 110
  Follow-up Visit Day 90 | 0

15. Primary Outcome: Change in Physician's Withdrawal Checklist (PWC-20) Total Score From Last Day on Treatment
Description: The PWC-20 is a rater-administered 20-item scale to assess signs and symptoms of withdrawal. Twenty items are rated on a 4-point scale as not present (0 points), mild (1 point), moderate (2 points), or severe (3 points). The points from all items are calculated as a total score. Higher scores indicate more severe withdrawal symptoms.
Time Frame: 1, 4, 7, 14, 21, and 90 days post last dose.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Change in Score on a Scale
Arm/Group | Combined Parent Treatment Group
Number analyzed (Participants) | 95
Change in Score on a Scale
  End of Treatment: number analyzed (Participants) | 72
  End of Treatment | -0.1 (6.33)
  Follow-up Visit Day 1: number analyzed (Participants) | 92
  Follow-up Visit Day 1 | -0.6 (5.06)
  Follow-up Visit Day 4: number analyzed (Participants) | 92
  Follow-up Visit Day 4 | -0.5 (4.51)
  Follow-up Visit Day 7 | -1.1 (4.33)
  Follow-up Visit Day 14: number analyzed (Participants) | 90
  Follow-up Visit Day 14 | -0.4 (4.93)
  Follow-up Visit Day 21: number analyzed (Participants) | 91
  Follow-up Visit Day 21 | -1.2 (5.31)
  Follow-up Visit Day 90 | -0.7 (5.15)

16. Primary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Score From Last Day on Treatment
Description: The HADS is a validated patient reported outcome for assessing anxiety and depression. It consists of 14 items in total, 7 items related to anxiety and 7 items related to depression. For each item patients select a statement (valued at 0 to 3 points) that closest matches their own feeling over the past week. Separate total scores for anxiety and depression are derived by adding up points. Total scores can range from 0 to 21 points. Higher scores indicate more severe anxiety and depression and scores of 8 to 10 are generally considered indicative of borderline anxiety/depression disorders and scores of 11 and higher are generally considered indicative of anxiety/depression disorders.
Time Frame: 1, 4, 7, 14, 21, and 90 days post last dose.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Change in Score on a Scale
Arm/Group | Combined Parent Treatment Group
Number analyzed (Participants) | 96
Change in Score on a Scale
  Depression - End of Treatment: number analyzed (Participants) | 72
  Depression - End of Treatment | 0.3 (3.17)
  Depression - Follow-up Visit Day 1: number analyzed (Participants) | 93
  Depression - Follow-up Visit Day 1 | -0.1 (2.15)
  Depression - Follow-up Visit Day 4: number analyzed (Participants) | 94
  Depression - Follow-up Visit Day 4 | -0.1 (2.13)
  Depression - Follow-up Visit Day 7: number analyzed (Participants) | 95
  Depression - Follow-up Visit Day 7 | -0.2 (2.29)
  Depression - Follow-up Visit Day 14: number analyzed (Participants) | 91
  Depression - Follow-up Visit Day 14 | 0.1 (2.36)
  Depression - Follow-up Visit Day 21: number analyzed (Participants) | 93
  Depression - Follow-up Visit Day 21 | 0.1 (2.35)
  Depression - 90-Day Safety Follow-up Visit | -0.2 (2.86)
  Anxiety - End of Treatment: number analyzed (Participants) | 72
  Anxiety - End of Treatment | -0.3 (2.76)
  Anxiety - Follow-up Visit Day 1: number analyzed (Participants) | 93
  Anxiety - Follow-up Visit Day 1 | -0.5 (2.33)
  Anxiety - Follow-up Visit Day 4: number analyzed (Participants) | 94
  Anxiety - Follow-up Visit Day 4 | -0.4 (2.30)
  Anxiety - Follow-up Visit Day 7: number analyzed (Participants) | 95
  Anxiety - Follow-up Visit Day 7 | -0.8 (2.47)
  Anxiety - Follow-up Visit Day 14: number analyzed (Participants) | 91
  Anxiety - Follow-up Visit Day 14 | -0.6 (2.17)
  Anxiety - Follow-up Visit Day 21: number analyzed (Participants) | 93
  Anxiety - Follow-up Visit Day 21 | -0.7 (2.35)
  Anxiety - 90-Day Safety Follow-up Visit | -0.7 (2.99)

17. Primary Outcome: Changes in Epworth Sleepiness Scale (ESS) Score From Last Day on Treatment
Description: The ESS is a validated self administered questionnaire with 8 questions. Respondents rate on a 4-point scale (0 to 3) their chances of dozing off or falling asleep while engaged in 8 different activities. The ESS score is the sum of 8 item scores and can range from 0 to 24 points. Higher scores indicate more daytime sleepiness.
Time Frame: 1, 4, 7, 14, 21, and 90 days post last dose.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Change in Score on a Scale
Arm/Group | Combined Parent Treatment Group
Number analyzed (Participants) | 96
Change in Score on a Scale
  End of Treatment: number analyzed (Participants) | 73
  End of Treatment | 0.4 (4.92)
  Follow-up Visit Day 1: number analyzed (Participants) | 93
  Follow-up Visit Day 1 | -0.6 (4.28)
  Follow-up Visit Day 4: number analyzed (Participants) | 94
  Follow-up Visit Day 4 | -0.5 (4.38)
  Follow-up Visit Day 7: number analyzed (Participants) | 95
  Follow-up Visit Day 7 | -0.7 (4.25)
  Follow-up Visit Day 14: number analyzed (Participants) | 92
  Follow-up Visit Day 14 | -0.9 (4.10)
  Follow-up Visit Day 21: number analyzed (Participants) | 93
  Follow-up Visit Day 21 | -0.9 (4.42)
  Follow-up Visit Day 90 | -0.8 (3.75)

18. Primary Outcome: Changes in Vital Sign Values From Last Day on Treatment
Description: Vital signs included sitting systolic blood pressure (SBP), sitting diastolic blood pressure (DBP).
Time Frame: 1, 4, 7, 14, 21, 28, and 90 days post last dose.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combined Parent Treatment Group
Number analyzed (Participants) | 252
mmHg
  Systolic Blood Pressure(mmHg)-Sitting: End of Treatment | -1.77 (11.189)
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 1: number analyzed (Participants) | 49
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 1 | 0.63 (8.311)
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 4: number analyzed (Participants) | 52
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 4 | -0.04 (8.931)
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 7: number analyzed (Participants) | 51
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 7 | 0.82 (7.911)
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 14: number analyzed (Participants) | 68
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 14 | -0.4 (8.128)
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 21: number analyzed (Participants) | 55
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 21 | 1.25 (9.029)
  Systolic Blood Pressure(mmHg)-Sitting: Safety Follow-up Visit -Day 28: number analyzed (Participants) | 213
  Systolic Blood Pressure(mmHg)-Sitting: Safety Follow-up Visit -Day 28 | -0.72 (11.135)
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 90: number analyzed (Participants) | 96
  Systolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 90 | -0.69 (10.865)
  Diastolic Blood Pressure(mmHg)-Sitting: End of Treatment | -1.10 (8.356)
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 1: number analyzed (Participants) | 49
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 1 | -1.18 (8.218)
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 4: number analyzed (Participants) | 52
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 4 | -2.02 (7.760)
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 7: number analyzed (Participants) | 51
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 7 | -1.80 (7.275)
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 14: number analyzed (Participants) | 68
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 14 | -1.82 (7.643)
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 21: number analyzed (Participants) | 55
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 21 | -1.00 (8.181)
  Diastolic Blood Pressure(mmHg)-Sitting: Safety Follow-up Visit -Day 28: number analyzed (Participants) | 213
  Diastolic Blood Pressure(mmHg)-Sitting: Safety Follow-up Visit -Day 28 | -1.21 (8.103)
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 90: number analyzed (Participants) | 96
  Diastolic Blood Pressure(mmHg)-Sitting: Follow-up Visit Day 90 | -2.01 (7.689)

19. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: The Annualized Relapse Rate (ARR) is the average number of relapses per study arm in one year. A relapse is defined as the occurrence of new or worsening neurological symptoms attributable to multiple sclerosis (MS) and immediately preceded by a relatively stable or improving neurological state of at least 30 days. The adjusted ARR was based on the negative binomial regression model with parent treatment group, adjusted for region (Eastern Europe vs Rest of World), age at parent baseline, and the parent baseline number of gadolinium-enhanced (GdE) lesions. The natural log transformation of time on treatment was used as an offset term to adjust for participants having different exposure times.
Time Frame: From first dose up until last dose of study treatment or data-cutoff date, whichever occurred first (up to approximately 87 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Proportion of participants | 0.097 [0.078 to 0.121] | 0.108 [0.088 to 0.133] | 0.090 [0.073 to 0.111]

20. Secondary Outcome: Time to First Relapse (TFR)
Description: The time between first dose of study treatment and first relapse if experienced by a participant. A participant was censored if follow-up ended before a relapse occurred, whether due to the participant completing study, withdrawing from the study, or due to the cutoff of data collection for the analysis. The censor date was the date of the end of study or the date of the data cutoff for participant who were ongoing. Participants who withdrew from the study after the baseline visit were censored at the last known date while on study. Based on Kaplan-Meier product limit estimates.
Time Frame: Overall: From first dose to first relapse, last dose, or data-cutoff date, whichever occurred first (up to approx 87 months); Visits: 2 weeks post first dose, 3 months post first dose, and every 3 months thereafter up until 81 months post first dose.
Population: All treated participants with confirmed relapse.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 223 | 272 | 276
Days | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events. | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events. | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events.

21. Secondary Outcome: Number of Participants Who Were Relapse Free
Description: The number of participants who did not experience relapse. A relapse is defined as the occurrence of new or worsening neurological symptoms attributable to multiple sclerosis (MS) and immediately preceded by a relatively stable or improving neurological state of at least 30 days.
Time Frame: From first dose to last dose of study treatment or data-cutoff date, whichever occurred first (up to approximately 87 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 736 | 877 | 881
Participants | 513 | 605 | 605

22. Secondary Outcome: Average Number of New or Enlarging Hyperintense T2-Weighted Brain MRI Lesions Per Scan at Each Visit
Description: Adjusted Mean of new enlarging T2 lesions per scan at each visit. Based on a negative binomial regression model, adjusted for parent study, region (Eastern Europe vs. Rest of the World), age at Baseline, and baseline number of GdE lesions.
  T2 Magnetic Resonance Imaging (MRI) sequences are used to highlight areas of demyelination in brain neurons, which happens when the outer layer of the neurons is damaged due to multiple sclerosis (MS) activity. T2 sequences can be used to count the total number of MS lesions, which look like bright white spots on T2 sequences, and can be called "hyperintense".
Time Frame: At 12 months post first dose and every 12 months thereafter up until 72 months post first dose.
Population: All treated participants with at least one on treatment MRI assessment showing new or enlarging lesions.
Measure: Mean (95% Confidence Interval); unit: New or Enlarging Lesions per Scan
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 696 | 722 | 726
New or Enlarging Lesions per Scan
  Month 12 | 1.532 [1.309 to 1.792] | 1.163 [0.995 to 1.360] | 1.302 [1.116 to 1.519]
  Month 24: number analyzed (Participants) | 651 | 683 | 698
  Month 24 | 1.254 [1.072 to 1.466] | 1.005 [0.862 to 1.172] | 1.190 [1.022 to 1.385]
  Month 36: number analyzed (Participants) | 605 | 643 | 655
  Month 36 | 1.136 [0.963 to 1.340] | 1.021 [0.872 to 1.197] | 1.142 [0.976 to 1.335]
  Month 48: number analyzed (Participants) | 570 | 585 | 591
  Month 48 | 0.935 [0.786 to 1.112] | 0.915 [0.770 to 1.087] | 1.044 [0.883 to 1.234]
  Month 60: number analyzed (Participants) | 527 | 575 | 565
  Month 60 | 0.791 [0.661 to 0.948] | 0.864 [0.728 to 1.025] | 0.935 [0.787 to 1.110]
  Month 72: number analyzed (Participants) | 136 | 162 | 164
  Month 72 | 0.800 [0.566 to 1.132] | 0.780 [0.567 to 1.074] | 0.926 [0.684 to 1.255]

23. Secondary Outcome: Average Number of Gadolinium-Enhanced (GdE) Brain MRI Lesions Per Scan at Each Visit
Description: Number of gadolinium-enhanced (GdE) (also called GdE enhanced T1) brain MRI lesions per scan at each visit.
  Increased numbers of GdE lesions indicates an increase in the in the amount of active inflammation at the site and may be indicative of progressive disease.
  Based on a negative binomial regression model, adjusted for parent study, region (Eastern Europe vs. Rest of the World), age at Baseline, and Baseline number of GdE lesions.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 72 months post first dose.
Population: All treated participants with baseline and at least one on treatment MRI assessment showing the presence of GdE brain MRI lesions.
Measure: Mean (95% Confidence Interval); unit: New or Enlarging Lesions
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 740 | 756 | 760
New or Enlarging Lesions
  Baseline | 0.460 [0.369 to 0.573] | 0.244 [0.193 to 0.308] | 0.177 [0.138 to 0.226]
  Month 12: number analyzed (Participants) | 695 | 723 | 725
  Month 12 | 0.106 [0.076 to 0.147] | 0.130 [0.097 to 0.175] | 0.205 [0.155 to 0.273]
  Month 24: number analyzed (Participants) | 651 | 683 | 698
  Month 24 | 0.138 [0.099 to 0.192] | 0.149 [0.109 to 0.205] | 0.224 [0.166 to 0.302]
  Month 36: number analyzed (Participants) | 604 | 642 | 653
  Month 36 | 0.194 [0.134 to 0.281] | 0.155 [0.109 to 0.221] | 0.243 [0.173 to 0.342]
  Month 48: number analyzed (Participants) | 569 | 584 | 590
  Month 48 | 0.230 [0.163 to 0.325] | 0.161 [0.108 to 0.241] | 0.245 [0.170 to 0.355]
  Month 60: number analyzed (Participants) | 525 | 576 | 565
  Month 60 | 0.074 [0.043 to 0.125] | 0.062 [0.037 to 0.104] | 0.076 [0.046 to 0.126]
  Month 72: number analyzed (Participants) | 136 | 161 | 164
  Month 72 | 0.099 [0.044 to 0.224] | 0.102 [0.049 to 0.213] | 0.082 [0.038 to 0.177]

24. Secondary Outcome: Time to Onset of Disability Progression as Defined by a Sustained Worsening in Expanded Disability Status Scale (EDSS)
Description: Multiple sclerosis (MS) disability progression is defined as a sustained worsening in EDSS of 1.0 points or more from baseline, confirmed after a 3-month and 6-month period. The EDSS is a standardized method, widely accepted, numerical scale used to evaluate disability in people with multiple sclerosis (MS). The EDSS is evaluated according to signs and symptoms observed during a standard neurological examination. These clinical observations are classified in 7 FS scales, each of them grading signs and symptoms for different neurological functions: pyramidal, cerebellar, brainstem, sensory, bowel or bladder, visual, and cerebral.
  Derived using Kaplan-Meier estimates.
Time Frame: At 3 and 6 months post first dose.
Population: All treated participants with disability progression data
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 122 | 160 | 146
Days
  Month 3 | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events. | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events. | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events.
  Month 6: number analyzed (Participants) | 116 | 135 | 128
  Month 6 | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events. | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events. | NA [NA to NA] — Median, UL and LL not estimable by KM methodology due to insufficient number of events.

25. Secondary Outcome: Number of Participants Free of Gadolinium-Enhanced (GdE) Brain Lesions at Each Visit
Description: Number of participants without gadolinium enhanced (GdE) brain MRI lesions at each visit. Increased numbers of GdE lesions indicates an increase in the in the amount of active inflammation at the site and may be indicative of progressive disease.
  Based on cumulative number of GdE lesions at a participant level.
Time Frame: At baseline and every 12 months thereafter up until 72 months post first dose.
Population: All participants in the intent to treat (ITT) population with baseline and at least one on treatment MRI assessment showing the absence of GdE brain lesions.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 740 | 756 | 760
Participants
  Baseline | 538 | 609 | 662
  Month 12: number analyzed (Participants) | 695 | 723 | 725
  Month 12 | 622 | 644 | 627
  Month 24: number analyzed (Participants) | 651 | 683 | 698
  Month 24 | 582 | 601 | 596
  Month 36: number analyzed (Participants) | 604 | 642 | 653
  Month 36 | 538 | 576 | 569
  Month 48: number analyzed (Participants) | 569 | 584 | 590
  Month 48 | 506 | 518 | 517
  Month 60: number analyzed (Participants) | 525 | 576 | 565
  Month 60 | 478 | 528 | 512
  Month 72: number analyzed (Participants) | 136 | 161 | 164
  Month 72 | 121 | 145 | 149

26. Secondary Outcome: Number of Participants Free of New or Enlarging T2 Lesions at Each Visit
Description: Number of participants without new or enlarging T2 brain MRI lesions at each visit. Some multiple Sclerosis (MS) lesions appear as bright spots in a T2-weighted MRI scan - these are called T2 lesions. The presence of new or larger T2 lesions may mean the participant is at higher risk of disability and may have a less favorable long-term outcome.
  Based on cumulative number of new or enlarging T2 lesions at a participant level.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 72 months post first dose.
Population: All participants in the intent to treat population with baseline and at least one on treatment MRI assessment for T2 hyperintense lesions.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 696 | 722 | 726
Participants
  Month 12 | 322 | 400 | 419
  Month 24: number analyzed (Participants) | 651 | 683 | 698
  Month 24 | 260 | 323 | 338
  Month 36: number analyzed (Participants) | 605 | 643 | 655
  Month 36 | 220 | 264 | 271
  Month 48: number analyzed (Participants) | 570 | 585 | 591
  Month 48 | 204 | 223 | 223
  Month 60: number analyzed (Participants) | 527 | 575 | 565
  Month 60 | 177 | 213 | 209
  Month 72: number analyzed (Participants) | 136 | 162 | 164
  Month 72 | 53 | 59 | 57

27. Secondary Outcome: Percent Change in Normalized Brain Volume (Atrophy) on Brain MRI Scans From Baseline at Each Visit
Description: Percent change in normalized brain volume (Atrophy) on brain MRI scans from baseline at each visit. Brain atrophy can be seen in the earliest stages of multiple sclerosis (MS) and is a reliable predictor of future physical and cognitive disability.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until approximately 87 months post first dose.
Population: All treated participants with baseline and at least one on treatment MRI assessment.
Measure: Mean (Standard Deviation); unit: Percent Volume Change from Baseline
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 596 | 611 | 623
Percent Volume Change from Baseline
  Month 12: number analyzed (Participants) | 558 | 573 | 569
  Month 12 | -0.407 (0.731) | -0.359 (0.607) | -0.385 (0.602)
  Month 24: number analyzed (Participants) | 480 | 506 | 515
  Month 24 | -0.702 (0.809) | -0.657 (0.713) | -0.671 (0.706)
  Month 36: number analyzed (Participants) | 410 | 443 | 454
  Month 36 | -0.992 (0.882) | -0.947 (0.825) | -0.977 (0.764)
  Month 48: number analyzed (Participants) | 392 | 406 | 416
  Month 48 | -1.241 (1.012) | -1.214 (0.980) | -1.233 (0.949)
  Month 60: number analyzed (Participants) | 341 | 361 | 375
  Month 60 | -1.485 (1.079) | -1.478 (1.014) | -1.544 (1.017)
  Month 72: number analyzed (Participants) | 69 | 89 | 103
  Month 72 | -1.889 (1.288) | -1.696 (1.118) | -1.922 (1.290)
  End of Treatment | -1.283 (1.206) | -1.298 (1.133) | -1.355 (1.121)

28. Secondary Outcome: Change in Multiple Sclerosis Functional Composite (MSFC) Score From Baseline at Each Applicable Visit
Description: The Multiple Sclerosis Functional Composite (MSFC) is a 3-part tool to measure disability progression in those with multiple sclerosis (MS). It assesses leg, arm, hand, and cognitive function using 3 individual scales: - The Timed 25-Foot Walk: To measure leg function - The 9-Hole Peg Test: To measure arm and hand function - The Symbol Digit Modalities Test (SDMT): To measure cognitive processing speed, flexibility, and calculation ability. Scores from each of the three are converted into Z-scores and averaged to create an overall composite score. The Low-Contrast Letter Acuity Test (LCLA) is performed with the MSFC using a set of charts to assess low contrast visual acuity. Each chart corresponds to a different contrast level, and charts are scored based on the number of letters identified correctly. A Z-score of 0 represents the population mean. Standard deviations above the mean represent a better outcome. Baseline refers to assessments on or before receiving study treatment.
Time Frame: At baseline and every 12 months thereafter up until 84 months post first dose.
Population: All treated participants with baseline and non-baseline MSFC Z-score assessments for the respective visit
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 702 | 721 | 732
Z-Score
  MSFC Z Score Month 12 | 0.058 (2.540) | -0.085 (0.488) | -0.064 (0.618)
  MSFC Z Score Month 24: number analyzed (Participants) | 679 | 695 | 711
  MSFC Z Score Month 24 | -0.072 (0.855) | -0.082 (0.615) | -0.086 (0.632)
  MSFC Z Score Month 36: number analyzed (Participants) | 636 | 666 | 677
  MSFC Z Score Month 36 | -0.105 (0.876) | -0.100 (0.529) | -0.109 (0.656)
  MSFC Z Score Month 48: number analyzed (Participants) | 594 | 630 | 633
  MSFC Z Score Month 48 | -0.162 (1.025) | -0.148 (0.611) | -0.103 (1.460)
  MSFC Z Score Month 60: number analyzed (Participants) | 573 | 605 | 609
  MSFC Z Score Month 60 | -0.182 (1.062) | -0.174 (0.675) | -0.148 (0.580)
  MSFC Z Score Month 72: number analyzed (Participants) | 433 | 462 | 483
  MSFC Z Score Month 72 | -0.248 (1.256) | -0.239 (0.745) | -0.219 (0.672)
  MSFC Z Score Month 84: number analyzed (Participants) | 0 | 1 | 0
  MSFC Z Score Month 84 |  | -0.099 (NA) — Insufficient number of assessments to calculate SD |
  MSFC Z Score (LCLA) Month 12: number analyzed (Participants) | 693 | 709 | 721
  MSFC Z Score (LCLA) Month 12 | 0.043 (1.919) | -0.059 (0.402) | -0.055 (0.483)
  MSFC Z Score (LCLA) Month 24: number analyzed (Participants) | 668 | 680 | 705
  MSFC Z Score (LCLA) Month 24 | -0.056 (0.655) | -0.064 (0.483) | -0.074 (0.509)
  MSFC Z Score (LCLA) Month 36: number analyzed (Participants) | 621 | 649 | 670
  MSFC Z Score (LCLA) Month 36 | -0.097 (0.686) | -0.089 (0.447) | -0.103 (0.542)
  MSFC Z Score (LCLA) Month 48: number analyzed (Participants) | 583 | 619 | 627
  MSFC Z Score (LCLA) Month 48 | -0.158 (0.796) | -0.149 (0.525) | -0.103 (1.125)
  MSFC Z Score (LCLA) Month 60: number analyzed (Participants) | 566 | 595 | 605
  MSFC Z Score (LCLA) Month 60 | -0.175 (0.837) | -0.181 (0.572) | -0.153 (0.505)
  MSFC Z Score (LCLA) Month 72: number analyzed (Participants) | 424 | 454 | 477
  MSFC Z Score (LCLA) Month 72 | -0.237 (0.983) | -0.250 (0.624) | -0.213 (0.590)
  MSFC Z Score (LCLA) Month 84: number analyzed (Participants) | 0 | 1 | 0
  MSFC Z Score (LCLA) Month 84 |  | -0.103 (NA) — Insufficient number assessments to calculate SD |

29. Secondary Outcome: Change in Multiple Sclerosis Quality of Life 54 Score From Baseline at Each Applicable Visit
Description: The Multiple Sclerosis Quality of Life 54 (MSQOL-54) questionnaire is a health-related quality of life (HRQOL) instrument specific for multiple sclerosis (MS). This 54-item instrument generates 12 subscales along with two summary scores (physical health and mental health - derived from a weighted combination of scale scores), and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The MSQOL-54 items are transformed to 0-100 scores, and final scores are obtained by averaging items within the scales. The overall quality of life is assessed in question 54, which is scored on a scale of 0-100. Higher scores indicate better health-related quality of life. Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 84 months post first dose.
Population: All treated participants with baseline and non-baseline MSQOL-54 scores for the respective visit
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 659 | 678 | 678
Scores on a Scale
  Month 12: number analyzed (Participants) | 653 | 678 | 678
  Month 12 | 0.1 (10.68) | -0.1 (10.55) | 0.2 (9.85)
  Month 24: number analyzed (Participants) | 659 | 677 | 678
  Month 24 | 0.8 (11.51) | -0.6 (10.76) | -0.3 (11.25)
  Month 36: number analyzed (Participants) | 622 | 650 | 649
  Month 36 | 0.1 (12.20) | -0.6 (11.23) | -0.4 (12.37)
  Month 48: number analyzed (Participants) | 585 | 613 | 609
  Month 48 | -0.3 (12.60) | -1.4 (12.66) | -1.4 (12.71)
  Month 60: number analyzed (Participants) | 553 | 595 | 582
  Month 60 | -1.1 (13.27) | -2.7 (13.11) | -2.1 (12.62)
  Month 72: number analyzed (Participants) | 445 | 478 | 478
  Month 72 | -1.6 (14.97) | -3.0 (13.42) | -3.0 (13.88)
  Month 84: number analyzed (Participants) | 0 | 1 | 0
  Month 84 |  | -0.3 (NA) — Insufficient number assessments to calculate SD |

30. Secondary Outcome: Change From Baseline in Volume of Gadolinium Enhanced T1 Lesions
Description: Change from baseline in volume of gadolinium enhanced T1 lesions. T1-lesions are permanently damaged areas of the brain that appear as dark spots or "black holes" on a type of MRI scan. The growth of T1 lesions may mean the participant's Multiple Sclerosis (MS) is progressing.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 72 months post first dose.
Population: All treated participants with baseline and at least one on treatment MRI assessment showing the presence of brain MRI lesions.
Measure: Mean (Standard Deviation); unit: Volume (cm^3) Change from Baseline
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 695 | 723 | 725
Volume (cm^3) Change from Baseline
  Month 12 | -0.092 (0.435) | -0.015 (0.229) | -0.004 (0.180)
  Month 24: number analyzed (Participants) | 651 | 683 | 698
  Month 24 | -0.099 (0.431) | -0.017 (0.193) | 0.009 (0.264)
  Month 36: number analyzed (Participants) | 604 | 642 | 653
  Month 36 | -0.089 (0.485) | -0.018 (0.183) | 0.012 (0.237)
  Month 48: number analyzed (Participants) | 569 | 584 | 590
  Month 48 | -0.081 (0.467) | -0.012 (0.204) | 0.017 (0.252)
  Month 60: number analyzed (Participants) | 525 | 576 | 565
  Month 60 | -0.090 (0.448) | -0.017 (0.217) | 0.000 (0.189)
  Month 72: number analyzed (Participants) | 136 | 161 | 164
  Month 72 | -0.044 (0.145) | 0.003 (0.157) | 0.014 (0.307)

31. Secondary Outcome: Change From Baseline in Volume of T2 Lesions
Description: Some multiple Sclerosis (MS) lesions appear as bright spots in a T2-weighted MRI scan - these are called T2 lesions. Larger T2 lesions may mean the participant is at higher risk of disability and may have a less favorable long-term outcome.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 72 months post first dose.
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Volume (cm^3) Change from Baseline
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 696 | 723 | 726
Volume (cm^3) Change from Baseline
  Month 12 | 0.190 (1.498) | 0.174 (1.154) | 0.278 (1.384)
  Month 24: number analyzed (Participants) | 651 | 683 | 698
  Month 24 | 0.307 (1.633) | 0.303 (1.503) | 0.518 (2.294)
  Month 36: number analyzed (Participants) | 605 | 643 | 655
  Month 36 | 0.536 (2.218) | 0.456 (1.597) | 0.711 (2.540)
  Month 48: number analyzed (Participants) | 570 | 585 | 591
  Month 48 | 0.695 (2.805) | 0.583 (1.975) | 0.952 (2.945)
  Month 60: number analyzed (Participants) | 527 | 575 | 565
  Month 60 | 0.709 (2.907) | 0.683 (2.470) | 0.987 (3.197)
  Month 72: number analyzed (Participants) | 136 | 162 | 164
  Month 72 | 0.889 (2.760) | 0.557 (2.465) | 1.234 (4.307)

32. Secondary Outcome: Change From Baseline in Volume of Unenhancing T1 Lesions
Description: Change from baseline in volume of unenhancing T1 lesions. T1-lesions are permanently damaged areas of the brain that appear as dark spots or "black holes" on a type of MRI scan. The growth of T1 lesions may mean the participant's Multiple Sclerosis (MS) is progressing.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 72 months post first dose.
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Volume (cm^3) Change from Baseline
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 695 | 723 | 726
Volume (cm^3) Change from Baseline
  Month 12 | -0.625 (2.012) | -0.772 (1.792) | -0.760 (1.869)
  Month 24: number analyzed (Participants) | 651 | 683 | 698
  Month 24 | -0.192 (1.837) | -0.465 (1.735) | -0.455 (1.758)
  Month 36: number analyzed (Participants) | 604 | 643 | 653
  Month 36 | -0.482 (2.913) | -0.618 (2.430) | -0.583 (2.249)
  Month 48: number analyzed (Participants) | 569 | 584 | 590
  Month 48 | -0.398 (3.025) | -0.423 (2.439) | -0.403 (2.171)
  Month 60: number analyzed (Participants) | 526 | 575 | 565
  Month 60 | -0.261 (2.885) | -0.356 (2.679) | -0.209 (2.134)
  Month 72: number analyzed (Participants) | 136 | 161 | 164
  Month 72 | -0.047 (2.209) | -0.372 (3.257) | -0.256 (2.036)

33. Secondary Outcome: Cumulative Number of New Unenhancing T1 Lesions
Description: Number of new unenhancing T1 lesions. T1-lesions are permanently damaged areas of the brain that appear as dark spots or "black holes" on a type of MRI scan. The appearance of new T1 lesions may mean the participant's MS is progressing.
  Derived as the cumulative number of new or enlarging T1 lesions relative to baseline at a participant level.
  Baseline refers to assessments made on or before the first day participants received study treatment.
Time Frame: At baseline and every 12 months thereafter up until 72 months post first dose.
Population: All treated participants with baseline and at least one on treatment MRI assessment showing new or enlarging lesions.
Measure: Mean (Standard Deviation); unit: New or Enlarging Lesions.
Arm/Group | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
Number analyzed (Participants) | 695 | 722 | 725
New or Enlarging Lesions.
  Month 12 | 1.9 (4.66) | 1.1 (2.86) | 1.2 (3.16)
  Month 24: number analyzed (Participants) | 651 | 683 | 697
  Month 24 | 2.7 (6.30) | 1.8 (5.04) | 2.2 (5.24)
  Month 36: number analyzed (Participants) | 604 | 642 | 653
  Month 36 | 3.6 (8.41) | 2.5 (7.04) | 3.0 (7.55)
  Month 48: number analyzed (Participants) | 568 | 584 | 590
  Month 48 | 4.6 (11.02) | 3.3 (8.67) | 4.3 (10.56)
  Month 60: number analyzed (Participants) | 525 | 574 | 564
  Month 60 | 4.8 (11.43) | 3.9 (10.18) | 4.9 (12.39)
  Month 72: number analyzed (Participants) | 136 | 161 | 163
  Month 72 | 4.5 (10.11) | 3.2 (8.76) | 5.8 (16.55)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed from first dose until study completion (assessed up to approximately 87 months). SAEs and Other AEs were assessed from first dose to 90-days post last dose (an average of 65 months up to a max of 85 months).
Description: The placebo 0.5 mg, placebo 1 mg, IFN-B-1a and RPC1063 0.5 mg and 1 mg parent groups were used to represent All-Cause Mortality, Serious Adverse Events and Other (Not Serious) Adverse Events.
  Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Parent Treatment Group: Placebo for RPC1063 0.5 mg; Parent Treatment Group: Placebo for RPC1063 1 mg: Participants received a 7-day titration regimen of RPC1063 to reach the targeted dose of 1.0 mg which was taken by mouth once per day until the end of the trial or until the Sponsor discontinued the development program. Participants were instructed to take RPC1063 at approximately the same time each day with or without food.
Arm/Group | Parent Treatment Group: Placebo for RPC1063 0.5 mg | Parent Treatment Group: Placebo for RPC1063 1 mg | Parent Treatment Group IFN-B-1a 30 ug | Parent Treatment Group: RPC1063 0.5 mg | Parent Treatment Group: RPC1063 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35 | 6/736 | 5/840 | 5/846
Serious Adverse Events (participants affected / at risk) | 7/37 | 3/35 | 108/736 | 132/840 | 131/846
Other Adverse Events (participants affected / at risk) | 27/37 | 26/35 | 598/736 | 663/840 | 659/846
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parent Treatment Group: Placebo for RPC1063 0.5 mg (N=37) | Parent Treatment Group: Placebo for RPC1063 1 mg (N=35) | Parent Treatment Group IFN-B-1a 30 ug (N=736) | Parent Treatment Group: RPC1063 0.5 mg (N=840) | Parent Treatment Group: RPC1063 1.0 mg (N=846)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinoatrial block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Kidney duplex (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Sebaceous naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hyperadrenocorticism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Blepharal pigmentation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1
Choroiditis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Ranula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 1 | 0
Biliary polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 3
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Chronic hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Abdominal wall infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 3 | 4 | 2
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 4 | 8 | 7
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 4 | 6 | 10
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Chronic hepatitis B (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Echinococciasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Measles (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 2 | 7
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 4 | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Bursal fluid accumulation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Mandibular mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Angiomyxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Borderline serous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 3
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6 | 5 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 1
Encephalitis autoimmune (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Epilepsia partialis continua (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 3 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Noninfective encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Radicular pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 2 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 1 | 0
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Needle issue (Product Issues) | 0 | 0 | 0 | 0 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Kidney hypermobility (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 1
Breast dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Hydrosalpinx (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Perineal fistula (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Reproductive tract disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 2
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 1
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Miscarriage of partner (Social circumstances) | 0 | 0 | 0 | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Parent Treatment Group: Placebo for RPC1063 0.5 mg (N=37) | Parent Treatment Group: Placebo for RPC1063 1 mg (N=35) | Parent Treatment Group IFN-B-1a 30 ug (N=736) | Parent Treatment Group: RPC1063 0.5 mg (N=840) | Parent Treatment Group: RPC1063 1.0 mg (N=846)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 28 | 31 | 36
Lymphopenia (Blood and lymphatic system disorders) | 3 | 6 | 83 | 92 | 73
Palpitations (Cardiac disorders) | 0 | 2 | 6 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 13 | 15 | 12
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 21 | 37 | 25
Gastritis (Gastrointestinal disorders) | 1 | 2 | 15 | 17 | 11
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 8 | 9 | 7
Vomiting (Gastrointestinal disorders) | 1 | 3 | 5 | 8 | 7
Fatigue (General disorders) | 2 | 3 | 17 | 27 | 29
Immunisation reaction (Immune system disorders) | 0 | 2 | 5 | 9 | 6
Bronchitis (Infections and infestations) | 1 | 3 | 38 | 58 | 55
COVID-19 (Infections and infestations) | 8 | 7 | 116 | 130 | 136
Herpes zoster (Infections and infestations) | 2 | 2 | 13 | 17 | 12
Influenza (Infections and infestations) | 0 | 4 | 24 | 32 | 24
Nasopharyngitis (Infections and infestations) | 5 | 9 | 164 | 176 | 177
Pharyngitis (Infections and infestations) | 0 | 3 | 30 | 39 | 35
Respiratory tract infection (Infections and infestations) | 2 | 1 | 53 | 56 | 53
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 46 | 52 | 46
Sinusitis (Infections and infestations) | 1 | 0 | 37 | 33 | 30
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 99 | 101 | 97
Urinary tract infection (Infections and infestations) | 8 | 3 | 48 | 52 | 58
Viral infection (Infections and infestations) | 1 | 2 | 7 | 7 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 11 | 8 | 13
Alanine aminotransferase increased (Investigations) | 3 | 3 | 46 | 40 | 34
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 23 | 20 | 15
Blood cholesterol increased (Investigations) | 0 | 4 | 5 | 7 | 8
Blood triglycerides increased (Investigations) | 0 | 2 | 4 | 3 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 4 | 71 | 63 | 61
Low density lipoprotein increased (Investigations) | 0 | 2 | 1 | 3 | 4
Lymphocyte count decreased (Investigations) | 7 | 2 | 68 | 77 | 81
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 15 | 10 | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 3 | 32 | 36 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 43 | 53 | 61
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 72 | 81 | 71
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 26 | 29 | 32
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 6 | 8 | 12
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 11 | 8 | 6
Headache (Nervous system disorders) | 2 | 7 | 131 | 142 | 144
Muscle spasticity (Nervous system disorders) | 0 | 2 | 3 | 9 | 13
Paraesthesia (Nervous system disorders) | 1 | 2 | 12 | 10 | 20
Anxiety (Psychiatric disorders) | 0 | 4 | 28 | 26 | 29
Depression (Psychiatric disorders) | 0 | 2 | 38 | 45 | 41
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 2 | 6 | 3
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 6 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 18 | 32 | 30
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 5 | 7 | 5
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 6 | 4
Hypertension (Vascular disorders) | 5 | 2 | 76 | 81 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02576717/Prot_SAP_000.pdf